CLINICAL TRIAL: NCT03479788
Title: Sleep and Stent Study II - Rapid Eye Movement Related Obstructive Sleep Apnea in Diabetic Versus Non-Diabetic Patients Treated With Percutaneous Coronary Intervention
Brief Title: Rapid Eye Movement Related OSA in Diabetic Versus Non-Diabetic Patients Treated With PCI
Status: Completed | Type: Observational
Sponsor: National University of Singapore (Other)
Collaborators: National Heart Centre Singapore (Other)
Responsible Party: Principal Investigator, Chi-Hang Lee, Associate Professor, National University of Singapore
Other Study IDs: Sleep and Stent Study II
Record Dates: First submitted 2018-03-21; First posted 2018-03-27 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Obstructive Sleep Apnea; Diabetes Mellitus; Coronary Artery Disease
Keywords: sleep apnea, coronary artery, diabetes
MeSH Terms: conditions — Sleep Apnea, Obstructive; Diabetes Mellitus; Coronary Artery Disease; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DM: Observational study. NO intervention
- non-DM: Observational study. NO intervention

SUMMARY:
The primary objective of the Sleep and Stent II is to determine the prevalence of REM-OSA in DM versus non-DM patients undergoing clinically indicated PCI.

The secondary objectives are to investigate the association between REM-AHI and (1) cardiac arrhythmia based on ambulatory ECG monitoring, (2) excessive daytime sleepiness, and (3) glycemic control in patients with DM.

In addition, we will determine the prevalence of REM-OSA based on alternative definitions, including (a) overall AHI at least 5 with AHI REM/AHI NREM ratio at least 2; (b) overall AHI at least 5 with AHI REM/AHI NREM ratio at least 2 and with AHI NREM < 15; (c) overall AHI at least 5, AHI REM/AHI NREM ratio at least 2 and with AHI NREM < 8.

DETAILED DESCRIPTION:
The Sleep and Stent II is a cross-sectional study of patients who have undergone PCI for coronary artery disease. A total of 200 adult patients who have undergone clinically indicated PCI between 6 and 36 months ago are eligible. The study involves the 2 national heart centers and the Ng Teng Fong General Hospital in Singapore (3 centers in total). The National University Heart Center Singapore is the leading center and it is responsible for the overall study design and study conduct. The estimated duration of the Sleep and Stent II is 3 years (2018-2020).

All subjects and/or their legally authorized representative must provide written informed consent before any study-related procedure can be conducted. The patients will be divided into DM and non-DM groups, and the two groups will be matched for age, sex, and BMI. As a standard clinical practice in Singapore, patients who have undergone PCI will be followed up at the outpatient clinic for continuation of care. As such, the recruitment will be conducted at the outpatient clinic. All recruited patients will undergo an overnight polysomnography at the National University Health System Cardiosleep research laboratory.

All polysomnography studies will be conducted using a standardized level I diagnostic device (Embla RemLogic, Natus Medical Inc. Canada). Outputs recorded from the portable diagnostic device will be manually scored by an independent sleep technologist with Registered Polysomnographic Technologist credentials, blinded to the patients' clinical characteristics.

The primary measure of the polysomnography will be the AHI, quantified as the total number of apneas and hypopneas per hour of sleep. An apnea is defined as a 90% or greater decrease in airflow from the baseline value for at least 10 seconds. Apneas are further classified as obstructive or central based on the presence or absence, respectively, of respiratory-related chest wall movement. Hypopnea is defined as a 30-90% reduction in airflow from the baseline value lasting 10 seconds or more, in conjunction with ≥3% oxygen desaturation. The respiratory event scoring will be performed according to the American Academy of Sleep Medicine guidelines. For all patients the AHI during total sleep time, the AHI during REM (AHI-REM), and the AHI during non-REM sleep (AHI-NREM) will be calculated. REM OSA is defined in a variety of ways including AHI at least 5 withAHI-REM/AHI-NREM ratio at least 2; overall AHI at least 5 with AHI-REM/ AHI-NREM ratio at least 2 and with AHI-NREM less than 15; overall AHI at least 5, AHI-REM/AHI-NREM ratio at least 2 and with AHI-NREM less than 8.

ELIGIBILITY:
Inclusion Criteria:

Age >21 years old Have undergone clinically indicated PCI between 6 and 36 months ago

Exclusion Criteria:

Known OSA on treatment Clinical instability with admission for acute coronary syndrome, heart failure or stroke in the past 30 days Inability to give informed consent

Ages: 22 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone clinically indicated PCI between 6 and 36 months ago
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
REM OSA | 1 day
  The primary measure of the polysomnography will be the AHI, quantified as the total number of apneas and hypopneas per hour of sleep. An apnea is defined as a 90% or greater decrease in airflow from the baseline value for at least 10 seconds. Apneas are further classified as obstructive or central based on the presence or absence, respectively, of respiratory-related chest wall movement. Hypopnea is defined as a 30-90% reduction in airflow from the baseline value lasting 10 seconds or more, in conjunction with =3% oxygen desaturation. The respiratory event scoring will be performed according to the American Academy of Sleep Medicine guidelines. For all patients the AHI during total sleep time, the AHI during REM (AHI-REM), and the AHI during non-REM sleep (AHI-NREM) will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Lee Chi-Hang Ronald, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided